CLINICAL TRIAL: NCT03202654
Title: A Randomized, Double-Blind, Controlled, Crossover, Pilot Trial Comparing the Effects of Corn and Coconut Oils on Fasting Lipoprotein Lipids and Markers of Insulin Sensitivity and Inflammation in Men and Women
Brief Title: Effects of Corn and Coconut Oils on Lipoprotein Lipids, Insulin Sensitivity and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: ACH Food Companies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: MB-1703
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Healthy Men and Women
MeSH Terms: interventions — Corn Oil; Coconut Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corn Oil Intervention (Experimental): Study products delivering 4 tablespoons/day corn oil will be administered for 4-week treatment period.
  Interventions: Other: Corn Oil
- Coconut Oil Intervention (Active Comparator): Study products delivering 4 tablespoons/day coconut oil will be administered for 4-week treatment period.
  Interventions: Other: Coconut Oil

INTERVENTIONS:
Other: Corn Oil — 4 tablespoons/day of corn oil for 4-week treatment period.
  Arms: Corn Oil Intervention
Other: Coconut Oil — 4 tablespoons/day of coconut oil for 4-week treatment period.
  Arms: Coconut Oil Intervention

SUMMARY:
The objectives of this trial are to assess the effects of corn oil and coconut oil on low-density lipoprotein cholesterol (LDL-C) concentrations, and other aspects of the fasting lipoprotein lipid profile, as well as insulin sensitivity and an inflammatory marker, in men and women.

DETAILED DESCRIPTION:
This is a randomized, crossover, pilot study that includes two screening visits and two 4-week test periods, separated by a 3-week washout. Subjects will consume study products providing 4 tablespoons oil/day of either corn oil or coconut oil replacing the same amount of oil in the background diet. Subjects will otherwise be encouraged to follow their habitual diet during both treatment periods. They will receive diet instructions on the incorporation of food substitutions during the test periods to maintain habitual energy intake. Subjects will record daily study product intake and compliance in a Daily Log. An intravenous glucose tolerance test (IVGTT) will be completed at baseline and the end of each treatment period for evaluation of insulin sensitivity. Fasting blood samples will be collected for lipid profile and high-sensitivity C-reactive protein (hs-CRP) measurements at all visits. Assessments of vital signs and body weight, review of concomitant medication/supplement use and inclusion and exclusion criteria for relevant changes, and evaluation of adverse effects will be performed throughout the study. Compliance will be assessed using the Daily Log intake percentages as the primary source.

ELIGIBILITY:
Inclusion Criteria:

1. BMI of 18.5-34.9 kg/m2.
2. Fasting LDL-C level ≥115 mg/dL and <190 mg/dL, and TG level ≤375 mg/dL.
3. Judged to be in general good health on the basis of medical history and screening laboratory tests.

Exclusion Criteria:

1. Atherosclerotic cardiovascular disease including any of the following:

   clinical signs of atherosclerosis including peripheral arterial disease, abdominal aortic aneurysm, carotid artery disease [symptomatic (e.g., myocardial infarction, angina, transient ischemic attack or stroke of carotid origin) or >50% stenosis on angiography or ultrasound] or other forms of clinical atherosclerotic disease (e.g., renal artery disease).
2. History or presence of clinically important pulmonary (including uncontrolled asthma), endocrine (including type 1 or 2 diabetes mellitus), chronic inflammatory disease (including irritable bowel disease, lupus, rheumatoid arthritis), hepatic, renal, hematologic, immunologic, dermatologic, neurologic, psychiatric, or biliary disorders.
3. Known allergy, sensitivity, or intolerance to any ingredients in the study products.
4. Uncontrolled hypertension.
5. Recent history of cancer, except for non-melanoma skin cancer.
6. Recent change in body weight of ± 4.5 kg.
7. Recent use of any medications intended to alter the lipid profile [e.g., statins, bile acid sequestrants, cholesterol absorption inhibitor, fibrates, niacin (drug form), omega-3-ethyl ester drugs, or proprotein convertase subtilisin kexin type 9 inhibitors].
8. Recent use of any foods or dietary supplement that might alter lipid metabolism [e.g., omega-3 fatty acid supplements (e.g., flaxseed, fish or algal oils) or fortified foods, sterol/stanol products; dietary supplements (including Metamucil® or viscous fiber-containing supplement); red rice yeast supplements; garlic supplements; soy isoflavone supplements; niacin or its analogues at doses >400 mg/d].
9. Recent use of weight-loss drugs or programs or antibiotics.
10. Recent daily use of non-steroidal anti-inflammatory drugs (except low-dose aspirin) or unstable use of antihypertensive medication.
11. Recent use of medications that influence carbohydrate metabolism (e.g., adrenergic receptor blockers, diuretics, hypoglycemic medications, and/or systemic corticosteroids).
12. Pregnant, planning to be pregnant during the study period, lactating, or of childbearing potential and unwilling to commit to the use of a medically approved form of contraception throughout the study period.
13. Extreme dietary habits (e.g., vegan or very low carbohydrate diet).
14. Current or recent history for drug or alcohol abuse.
15. History of a diagnosed eating disorder (e.g., anorexia or bulimia nervosa).
16. Exposure to any non-registered drug product.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Percent change in LDL-C | Up to 28 days for each treatment period.
  Percent change in LDL-C from baseline (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 2-week and 4-week visits of each test period).

SECONDARY OUTCOMES:
Percent change in non-high-density lipoprotein cholesterol (Non-HDL-C). | Up to 28 days for each treatment period.
  Percent change in Non-HDL-C from baseline (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 2-week and 4-week visits of each test period).
Percent change in Total Cholesterol (TC) | Up to 28 days for each treatment period.
  Percent change in TC from baseline (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 2-week and 4-week visits of each test period).

OTHER OUTCOMES:
Percent change in Triglycerides (TG) | Up to 28 days for each treatment period.
  Percent change in TG from baseline (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 2-week and 4-week visits of each test period).
Percent change in high-density lipoprotein cholesterol (HDL-C). | Up to 28 days for each treatment period.
  Percent change in HDL-C from baseline (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 2-week and 4-week visits of each test period).
Percent change in TC/ (HDL-C) ratio. | Up to 28 days for each treatment period.
  Percent change in TC/ HDL-C ratio from baseline (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 2-week and 4-week visits of each test period).
Disposition index [acute insulin response to intravenous glucose (AIRg) x IV-SI] | Up to 50 minutes - measured at baseline, and end of each treatment period.
  Percent change (or change) from baseline to the end of each treatment period.
Glucose fractional disappearance rate from t = 10-50 min (Kg) | Up to 50 minutes - measured at baseline, and end of each treatment period.
  Percent change (or change) from baseline to the end of each treatment period.
Homeostasis model assessments of insulin sensitivity (HOMA%S) | Up to 28 days of each treatment period.
  Percent change or change from baseline to end of each treatment condition.
Beta-cell function (HOMA%B) | Up to 28 days of each treatment period.
  Percent change or change from baseline to end of each treatment condition.
Insulin sensitivity index (IV-SI) | Up to 50 minutes - measured at baseline, and end of each treatment period.
  Percent change or change from baseline to end of each treatment condition.
Percent change in high-sensitivity C-reactive protein (hs-CRP) | Up to 28 days for each treatment period.
  Percent change in hs-CRP from baseline (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 2-week and 4-week visits of each test period).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MB Clinical Research, Boca Raton, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois

REFERENCES:
- [Derived] Maki KC, Hasse W, Dicklin MR, Bell M, Buggia MA, Cassens ME, Eren F. Corn Oil Lowers Plasma Cholesterol Compared with Coconut Oil in Adults with Above-Desirable Levels of Cholesterol in a Randomized Crossover Trial. J Nutr. 2018 Oct 1;148(10):1556-1563. doi: 10.1093/jn/nxy156. PMID 30204921